CLINICAL TRIAL: NCT04556708
Title: Ozonated Water Irrigation as an Adjunct to Mechanical Periodontal Therapy in Patients With Periodontitis: A Randomized Clinical Trial
Brief Title: Ozonated Water Irrigation as an Adjunct to Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ozge Gokturk, Principal Investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-18
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Periodontal Diseases
Keywords: ozone; periodontitis; chlorhexidine digluconate; root planing
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline control group (Active Comparator): Periodontal clinical parameters and gingival crevicular fluid (GCF) samples were evaluated at baseline and 8 weeks after periodontal treatment in patients with periodontal disease.
  Intervention: Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with saline was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Interventions: Other: salin irrigation
- ozone group (Active Comparator): Periodontal clinical parameters and gingival crevicular fluid (GCF) samples were evaluated at baseline and 8 weeks after periodontal treatment in patients with periodontal disease.
  Intervention: Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with ozoned water was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Interventions: Other: ozonated water irrigation
- chlorhexidine group (Active Comparator): Periodontal clinical parameters and gingival crevicular fluid (GCF) samples were evaluated at baseline and 8 weeks after periodontal treatment in patients with periodontal disease.
  Intervention: Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with 0.12% chlorhexidine digluconate was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Interventions: Other: chlorhexidine irrigation

INTERVENTIONS:
Other: salin irrigation — Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with saline was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Arms: saline control group
Other: ozonated water irrigation — Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with ozonated water was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Arms: ozone group
Other: chlorhexidine irrigation — Non-surgical periodontal treatment (SRP and oral hygiene instructions) was performed and subgingival irrigation with 0.12% chlorhexidine digluconate was performed. Gingival crevicular fluid (GCF) samples were taken for vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) examination.
  Arms: chlorhexidine group

SUMMARY:
The use of chlorhexidine or ozonized water in periodontal pockets accompanying NPT can provide a significant improvement in probing pocket depths compared to conventional treatment. However, the effect of subgingival ozonized water applications on VEGF and IGF levels, which are thought to play a role in the pathogenesis of periodontal disease and periodontal regeneration, should be examined.

DETAILED DESCRIPTION:
Background: This study aims to evaluate the effects of subgingival ozonated water irrigation as an adjunct to non-surgical periodontal treatment on clinical and biochemical parameters of patients with moderate and severe periodontitis.

Methods: A total of 72 stage II and Stage III periodontitis patients were included in the study. The systemically healthy patients which were between the ages of 19 and 58 were treated non-surgically. At the end of each visit concerning periodontal treatment, the pocket of each tooth was irrigated with a sterile plastic syringe (10 mL per quadrant) with a blunt tip containing ozonated water (OW; ozone groups), 0.12% chlorhexidine digluconate (CHX groups) or saline (C; control groups) for 30-60 s. Periodontal clinical parameters, gingival crevicular fluid (GCF) vascular endothelial growth factor (VEGF) and insulin-like growth factor-1 (IGF-1) levels were evaluated at baseline and 8 weeks after periodontal treatment. All statistical data were analyzed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* good general health without a history of systemic disease (hyperthyroid, diabetes, etc.)
* ≥ 20 teeth
* having not received periodontal treatment within the past 6 months
* no contraindication for periodontal therapy and ozone application
* presenting moderate-to-severe periodontitis according to criteria outlined by 2017 World Workshop.

Exclusion Criteria:

* smoking
* use of anti-inflammatory and antibiotic drugs within the past 6 months
* pregnancy, lactation or use of oral contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
vascular endothelial growth factor level | Baseline and after 8 weeks
  Changes in the concentration of vascular endothelial growth factor in all groups within 8 weeks after periodontal treatment were measured.

SECONDARY OUTCOMES:
insulin-like growth factor-1 level | Baseline and after 8 weeks
  Changes in the concentration of insulin-like growth factor-1 in all groups within 8 weeks after periodontal treatment were measured.
Probing pocket depth | Baseline and after 8 weeks
  The changes in probing pocket depth before and after periodontal treatment were measured in 72 participants to determine the severity of disease and clinic outcome.
Clinical attachment level | Baseline and after 8 weeks
  The changes in clinical attachment level before and after periodontal treatment were measured in 72 participants to determine the severity of disease and clinic outcome.
Gingival index | Baseline and after 8 weeks
  The changes in gingival index level before and after periodontal treatment were measured in 72 participants to determine the severity of the disease.
Plaque index | Baseline and after 8 weeks
  The changes in gingival index level before and after periodontal treatment were measured in 72 participants to determine the severity of disease and clinic status.
Bleeding on probing | Baseline and after 8 weeks
  The changes in bleeding on probing before and after periodontal treatment were measured in 72 participants to record for classifying and evaluate (apically) gingival inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Gokturk, Principal Investigator — Abant Izzet Baysal
Locations (1):
- Abant Izzet Baysal, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No